CLINICAL TRIAL: NCT05222477
Title: Effect of Pelvic Floor Versus Abdominal Muscle Exercises on Nocturia and Sleep Quality in Women With Type 2 Diabetes
Brief Title: Abdominal Muscle Exercises on Nocturia and Sleep Quality in Women With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Principal Investigator, Hady Atef Labib, Lecturer of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NSQ
Record Dates: First submitted 2022-01-10; First posted 2022-02-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Nocturia; Sleep Deprivation
Keywords: nocturia; sleep deprivation; sleep quality; type 2 diabetes mellitus
MeSH Terms: conditions — Nocturia; Sleep Deprivation; Sleep Initiation and Maintenance Disorders; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic floor group (Active Comparator): pelvic floor exercises (intervention) will be applied for patients with nocturia and type 2 DM for 6 weeks, 3 times/week
  Interventions: Behavioral: pelvic floor exercise
- Abdominal group (Active Comparator): Abdominal exercises (intervention) will be applied for patients with nocturia and type 2 DM for 6 weeks, 3 times/week
  Interventions: Behavioral: Abdominal muscles exercise

INTERVENTIONS:
Behavioral: pelvic floor exercise — pelvic floor exercises(intervention) will be applied for patients with nocturia and type 2 DM for 6 weeks, 3 times/week
  Arms: Pelvic floor group
Behavioral: Abdominal muscles exercise — abdominal exercises (intervention) will be applied for patients with nocturia and type 2 DM for 6 weeks, 3 times/week
  Arms: Abdominal group

SUMMARY:
Nocturia is the leading cause of sleep disruption with its subsequent negative impact on general health and QoL for a large proportion of the adult population. Nocturia is prevalent in men and women of all ages but may be particularly bothersome in younger adults, in whom the consequences of sleep disturbance may be more detrimental for daytime functioning and possibly for health and mortality.The underlying causes of nocturia obviously influence the efficacy of different treatment options. Because a major cause of nocturia is overproduction of urine at night, nocturia may not respond to treatments designed to reduce urgency and increase bladder capacity or increase urine flow, such as agents for the management of bladder outlet obstruction.

DETAILED DESCRIPTION:
Nocturia may be more than simply a patient inconvenience, in view of its association with increased risk of morbidity and mortality. Clinicians often underestimate the consequences of nocturia, however, and thus fail to perform a thorough evaluation of the condition and its causes. Patients with nocturia deserve full consultation and implementation of an appropriate management strategy to ensure that the specific underlying medical conditions associated with nighttime voiding are addressed. Investigators should help women with nocturia as to improve their sleep. Participants will strengthen their pelvic floor muscles and abdominal muscles to control voiding so their sleep will not disturb to decrease their sufferance.

ELIGIBILITY:
Inclusion Criteria:

* Female Patients have had type II diabetes mellitus for more than 5years.
* HbA1c value from 6.5% to7.5%.
* Sleep deprivation for more than one month.
* Medically stable patients
* Blood glucose level from 130 to 150
* Patients are not pregnant
* Body mass index is 25 to 29.9 kg / m

Exclusion Criteria:

* Unstable medical condition.
* On antidepressors or anxiety treatment.
* With ant musculoskeletal or neurological conditions that might interfere with the execution or the assessment of the exercise.
* Cushing's disease (hypercortisolism) or Addison's disease (hypocortisolism).

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Nocturia is more prevalent in women with type 2 diabetes, therefore, we will include only females
Enrollment: 60 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Number of voids | 6 weeks
  Number of times that the patient go for toilet per night for urination
Sleep quality (0 is best, 3 is worst) | 6 weeks
  data about sleep from Pittsburgh sleep quality index questionnaire

SECONDARY OUTCOMES:
Abdominal and pelvic floor muscle electrical activity | 6 weeks
  Data described by the electromyograph (EMG)

CONTACTS AND LOCATIONS:
Overall Officials: Hady Atef, PhD, Principal Investigator — Cairo University
Locations (1):
- Alkasr Alaini hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
We are planning to share the IPD on publication
Supporting Information: Study Protocol
Time Frame: 12 months
Access Criteria: We will provide this to the journal where we will submit our manuscript